CLINICAL TRIAL: NCT05910268
Title: Innovations in Decentralizing HIV Services in Peru
Brief Title: Peru Decentralized HIV Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000035127; 1R01AI177082-01A1 (NIH)
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: HIV
Keywords: HIV Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Control (month 7-12) then NIATx+ECHO (month 13-36) then Maintenance (month 37-54)
  Interventions: Behavioral: NIATx + ECHO
- Group 2 (Experimental): Control (month 7-18) then NIATx+ECHO (month 19-42) then Maintenance (month 43-54)
  Interventions: Behavioral: NIATx + ECHO
- Group 3 (Experimental): Control (month 7-24 then NIATx+ECHO (month 25-48) then Maintenance (month 49-54)
  Interventions: Behavioral: NIATx + ECHO

INTERVENTIONS:
Behavioral: NIATx + ECHO — Project ECHO will be combined with NIATx to provide clinical skills to PHC staff and delivered in a hub and spoke model to connect SHC and PHC staff in delivery of HIV care. Decentralization will occur through guideline concordance, facilitated through NIATx and ECHO.

SUMMARY:
The purpose of this study is to understand the processes by which HIV care is decentralized, an evidence-informed strategy to improve retention in HIV care, in Peru. Decentralization of HIV services has not been evaluated using experimental designs and urban decentralization studies of HIV are uncommon, so this study will lend important insights for future decentralization efforts in Peru and other countries.

DETAILED DESCRIPTION:
Aim 1: Using the Delphi method, to create guidelines to identify: 1) criteria for transferring patients between hub and spoke and for initiating treatment in primary health clinics (PHCs); and 2) the most important quality health indicators (QHIs) needed to be assessed at PHCs to improve Retention in Care (RIC) and Viral Suppression (VS).

Aim 2: To identify the barriers and facilitators to decentralized HIV care from patients and clinicians in Secondary Health Centers (SHCs) and PHCs in Peru, where HIV is concentrated in key populations and treated primarily in SHCs. Findings will guide a hub and spoke decentralized care model to facilitate decentralized HIV care.

Aim 3: Using a step-wedge design with 4 hub/spokes (4 SHCs + 165 PHCs), the investigators will conduct a Type 2 hybrid implementation trial using to assess the extent to which decentralized services are adopted and scaled-up in PHCs over 24 months of observation using NIATx (Network for the Improvement of Addiction Treatment) combined with ECHO (Extension for Community Healthcare Outcomes)-like tele-education to develop and enhance a Hub and Spoke model. The implementation outcomes will include the proportionate increase of People with HIV (PWH): a) treated in PHCs; b) retained in care; and 3) achieving VS. Adoption by PHCs to accept PWH, fidelity to NIATx and ECHO, and concordance with decentralization guidelines will also be assessed.

The focus of this registration is Aim 3.

ELIGIBILITY:
Inclusion Criteria for Aim 3:

Survey of PHC and SHC Clinicians (N=330):

* Currently employed at a PHC or SHC that is participating in the study. Provide consent for participation.

Continuing Professional Development (N=825):

* Currently employed as a nurse or physician who fulfilled the ECHO training requirements

Survey of PHC Leadership (N=165):

* Currently serving as the leader of a PHC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1450 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of diagnosed PWH in treatment in PHC within the district | up to month 54
  The percentage of diagnosed PWH in treatment in PHC within the district will be used to assess the extent to which decentralized services are adopted and scaled-up in PHCs. Higher percentage indicates more services adopted and scaled-up.

SECONDARY OUTCOMES:
Effectiveness assessed as the extent of RIC and VS within the district | up to month 54
  The extent to which PWH are transferred from SHCs to PHCs and consequently are RIC and achieve VS assessed by the number of participants that are RIC and achieve VS

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Altice, M.D., M.A., Principal Investigator — Yale University
Locations (2):
- Yale University, New Haven, Connecticut, United States
- CITBM - Centro de Investigaciones Tecnológicas Biomédicas y Medioambientales, Bellavista, Peru

IPD SHARING:
Plan to Share IPD: Yes